CLINICAL TRIAL: NCT01995526
Title: A Single Dose Study to Evaluate the Pharmacokinetics and Glucodynamics of Insulin Peglispro (LY2605541) in Healthy Male Japanese Subjects
Brief Title: A Study of Insulin Peglispro in Healthy Male Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14682; I2R-JE-BIDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-11-21; First posted 2013-11-26 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — basal insulin peglispro; LY2605541

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Insulin Peglispro (Experimental): Single subcutaneous dose of 1.3 Units per kilogram (U/kg) insulin peglispro on Day 1.
  Interventions: Drug: Insulin Peglispro

INTERVENTIONS:
Drug: Insulin Peglispro
  Other Names: LY2605541

SUMMARY:
The main purpose of this study is to evaluate how the body processes the study drug known as insulin peglispro and how the study drug affects blood sugar in healthy male Japanese participants. This study will also evaluate safety of the study drug. The study will last up to 46 days for each participant, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Participants are overtly healthy male Japanese.
* Participants have Body Mass Index (BMI) between 18.5 and 25.0 kilograms per square meter (kg/m^2), inclusive.

Exclusion Criteria:

* Participants have known allergies to insulin peglispro or related compounds.
* Participants have a fasting venous blood glucose >108 milligrams per deciliter (mg/dL) (>6 millimoles per liter [mmol/L]).

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Peglispro
Started | 11
Received One Dose of Study Drug | 11
Completed | 10
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Insulin Peglispro: Single subcutaneous dose of 1.3 U/kg insulin peglispro on Day 1.
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.8 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 11
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 11

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Observed Maximum Concentration (Cmax) of Insulin Peglispro
Time Frame: Predose and 2, 4, 8, 12, 24, 30, 36, 48, 96, 144, and 192 hours postdose
Population: All participants who received insulin peglispro and had evaluable Cmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles/liter (pmol/L)
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 10
picomoles/liter (pmol/L) | 3720 (32)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of Insulin Peglispro
Description: AUC from time zero to infinity (AUC[0-∞]) of insulin peglispro was evaluated.
Time Frame: Predose and 2, 4, 8, 12, 24, 30, 36, 48, 96, 144, and 192 hours postdose
Population: All participants who received insulin peglispro and had evaluable AUC(0-∞) data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hours/liter (pmol*h/L)
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 10
picomoles*hours/liter (pmol*h/L) | 280000 (18)

3. Primary Outcome: Pharmacokinetics: Time of Maximum Observed Drug Concentration (Tmax) of Insulin Peglispro
Time Frame: Predose and 2, 4, 8, 12, 24, 30, 36, 48, 96, 144, and 192 hours postdose
Population: All participants who received insulin peglispro and had evaluable Tmax data.
Measure: Median (Full Range); unit: hours
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 10
hours | 39.00 [8.00 to 48.00]

4. Primary Outcome: Glucodynamics: Maximum Glucose Infusion Rate (Rmax)
Time Frame: Predose up to 36 hours post clamp procedure
Population: All participants who received insulin peglispro and had evaluable Rmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/minute/kilogram (mg/min/kg)
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 10
milligrams/minute/kilogram (mg/min/kg) | 1.75 (30)

5. Primary Outcome: Glucodynamics: Total Amount of Glucose Infused (Gtot)
Time Frame: Predose up to 36 hours post clamp procedure.
Population: All participants who received insulin peglispro and had evaluable Gtot data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilograms (mg/kg)
Arm/Group | Insulin Peglispro
Number analyzed (Participants) | 10
milligrams/kilograms (mg/kg) | 2180 (48)

ADVERSE EVENTS:
Arm/Group | Insulin Peglispro
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Peglispro (N=11)
Body temperature increased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days